CLINICAL TRIAL: NCT06309355
Title: A Randomized, Placebo-controlled, Double-blind, Multi Center, Phase IIa Trial Investigating the Safety, Tolerability, Pharmacokinetics and Efficacy of Topical Ointment YR001 in Adult Patients With Mild to Moderate Atopic Dermatitis
Brief Title: Topical YR001 Ointment in Adult With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hangzhou Yirui Pharmaceutical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YR001-A03
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis
Keywords: YR001; KV1.3
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active dose (Experimental): The intervention is YR001 ointment on a range of body surface area for multiple topical administration
  Interventions: Drug: YR001 ointment
- Placebo dose (Experimental): The intervention is Placebo on a range of body surface area for multiple topical administration
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: YR001 ointment — The intervention is YR001 ointment on a range of body surface area for multiple topical administration
  Arms: Active dose
Other: Placebo — The intervention is Placebo on a range of body surface area for multiple topical administration
  Arms: Placebo dose

SUMMARY:
This study is to evaluate the safety, tolerability, and pharmacokinetics of YR001 topical ointment in adult patients with mild to moderate atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the subject.
2. Male or female subject is aged 18 or older.
3. Subject has a weight of at least 50 kg and a body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive.
4. An Investigator Static Global Assessment (ISGA) score of 2 (mild) to 3 (moderate) at screening and Baseline.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Any skin tattoo, scar, cuts, bruises, or other skin damage, including excessive UV exposure, at the possible IP application sites.
3. Patients who have a source of itch solely or significantly from untreatable areas (face, scalp, genitals, palms of hands or soles of feet).
4. Have concomitant skin disease or infection (e.g., acne, impetigo) or presence of skin comorbidities in the skin areas to be dosed that may interfere with study assessments and treatment response.
5. Participation in another interventional clinical trial (e.g. investigational drug, biological agent, or device) within 30 days or 5 half-lives of investigational agent (whichever is longer) before entering, or during the trial, or previous participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be safety. Specifically, the primary endpoint will be the incidence of treatment-related AEs (TRAEs) through Day 50. | Day1-Day 50
  incidence of treatment related AEs (TRAEs)

SECONDARY OUTCOMES:
all treatment-emergents AEs | Day1-Day 50
  number, severity, causality, and outcome of all treatment-emergetns AEs (TEAEs)
Efficacy of YR001 Ointment | Day1-Day50
  Proportion of patients achieving ISGA 0 or 1 by visit

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Encore Medical Research -Boynton Beach, Boynton Beach, Florida
  - Encore Medical Research-Hollywood, Hollywood, Florida
  - Encore Medical Research-Weston, Weston, Florida
  - DelRicht Research, Baton Rouge, Louisiana

IPD SHARING:
Plan to Share IPD: No